CLINICAL TRIAL: NCT01122628
Title: Long Term Follow Up Study Into The Use Of The DVR-A Locking Plate In The Treatment Of Distal Radial Fractures
Brief Title: Long Term Follow up of the DVR-A Locking Plate
Status: Completed | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: DePuy International (Industry); Global Diagnostics UK (Other)
Responsible Party: Sponsor
Other Study IDs: 2009ORTH11; ISS2009050 (Other Grant/Funding Number: De Puy)
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Distal Radial Fractures Treated With a DVR-A Locking Plate
Keywords: Distal Radial Fracture; Volar Locking Plate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- DVR-A: Patients with a distal radial fracture treated with a DVR-A locking plate
  Interventions: Device: ORIF with DVR-A locking plate

INTERVENTIONS:
Device: ORIF with DVR-A locking plate — Size, length of plate and number os screws decided by operating surgeon
  Other Names: Distal volar radial anatomic plate; Hand inovations

SUMMARY:
The surgical treatment of wrist fractures (distal radius bone) has been changed by the introduction of a new plate design, the locking plate. This results in improved fixation and stabilisation of the fracture fragments allowing early movement.

This type of plate has been increasingly used throughout the world but questions have been raised regarding the potential complications of the surgery, particularly nerve and tendon injury. The Norfolk and Norwich Hospital has treated over 250 distal radial fractures with this type of plate. The investigators plan to recall these patients to asses their long term function, general satisfaction and radiological results.

ELIGIBILITY:
Inclusion Criteria:

* Treatment between Jan 2005 and March 2009

Exclusion Criteria:

* Under 16
* Unable to consent
* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be taken from a population consisting of all patients who have undergone distal radial fracture treatement with a DVR-A locking plate at the norfolk and Norwich University hospitals NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
DASH score | One year or more post surgery
  Disability of arm shoulder and hand score. This is a patient administered validated score
Pain | One year or more post surgery
  A patient administered visual analogue scale numbered 1-10. A mark can be placed anywhere along the line with a score of 0 indicating no pain and 10 the worst pain imaginable

SECONDARY OUTCOMES:
Complications | One year or more post surgery
  Examination and questioning by a hand therapist to pick up complications. Prompting for tendon irritation or rupture, neurovascular injury, plate or screw failure, hardware removal and infection
Radiographic appearance | One year or more post surgery
  Review of xrays to measure radial inclination, volar tilt,, shortening, articular stepoff and degenerative change
EQ 5D | More than one year post surgery
  Euroqual 5D is a patient administered general health questionaire that is validated.
Grip Strength | One year or more post surgery
  Measured by a dynomometer and referenced to the non operated side
Range of motion | One year or more post surgery
  Measured with a goniometer. Measurements taken of movements in the axial,coronal and sagital planes
Pain | One year or more post surgery
  A patient administered visual analogue scale numbered 1-10. A mark can be placed anywhere along the line with a score of 0 indicating no pain and 10 the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Adrian J Chojnowski, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom